CLINICAL TRIAL: NCT03466398
Title: Effects of a Remote Patient Monitoring Protocol on Glycemic Control in Adolescents With Type 1 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical limitations encountered with the remote monitoring platform
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Vivify Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STU 122016-056
Record Dates: First submitted 2018-02-20; First posted 2018-03-15 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Mellitus; Type 1 Diabetes Mellitus
Keywords: Remote Patient Monitoring; Adolescents
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Patients will use the Vivify Health RPM protocol as part of their diabetes management. They required to complete the Care Plan questions on a daily basis, and will upload blood glucose readings directly to the tablet twice a day. They will also have scheduled video conferences with study team physicians or advanced practice nurses on a weekly basis, to discuss ongoing diabetes management and educational objectives.
  Interventions: Behavioral: Vivify Health RPM Protocol
- Control Arm (No Intervention): Patients in this arm will manage their diabetes at home per normal standard of care, without any extra intervention from the study investigators.

INTERVENTIONS:
Behavioral: Vivify Health RPM Protocol — The Vivify RPM Protocol includes a wireless tablet and glucometer/Bluetooth device that can directly upload blood glucose readings to the tablet. Patients will daily Care Plan questionnaires on the tablet, as well as upload blood glucose readings twice a day. The tablets will also be used for weekly video conferences with study investigators.
  Arms: Intervention Arm

SUMMARY:
This study will use a randomized, crossover design. Children aged 13-18 years who have been diagnosed with Type 1 diabetes for at least 1 year and with at least 2 Hemoglobin A1c values ≥10.0% more than 60 days apart within the past year, with the most recent HbA1c value between 10-14%, will be placed into two separate treatment groups. Group A will undergo home monitoring for 12 weeks through the use of the Vivify kit, which contains a wireless tablet with daily medication/diet/symptom questionnaires. Group B will initially continue diabetes management per standard of care, including quarterly office visits. After a period of 12 weeks, Group B will switch to the RPM protocol, while Group A will return to standard of care. Both groups will have HbA1c values checked at the 0, 3, and 6 month time periods to assess the effect of the remote monitoring protocol. Participation in the RPM protocol will involve daily completion of the Care Plan questions, as well as weekly uploads of blood glucose values using the Glooko, Inc (Mountain View, CA) application, and weekly video visits with a member of the endocrinology team that will aim to address barriers to optimal care, whether they be motivation, knowledge or other difficulties. Barriers to care will be assessed in part through the completion of knowledge and self-efficacy assessments.

DETAILED DESCRIPTION:
RPM Software The Remote Patient Monitoring application that will be used for this study was created by Vivify Health. Vivify Health was founded in 2009, and their Remote Care Management platform utilizes consumer electronics and wireless health devices that patients can use easily from home. Using this platform, providers can create customized care plans for patients, as well as provide education through multimedia and face-to-face interaction through video conferences.

The Glooko mobile application allows patients to download diabetes data, including blood sugar readings, directly from their meter to compatible iOS and Android devices. The data can then be uploaded by the patient and viewed by providers.

Subjects Prospective study participants will be screened for by review of HbA1c values of patients with upcoming Endocrine clinic appointments, or during diabetes-related hospital admissions. Qualifying patients will be invited to participate in the study and written consent will be obtained from their parents (and assent from patients 10 years of age and older) prior to their randomization. Patients agreeing to participate in the study will be randomly assigned using sealed, blinded envelopes to Group A or Group B. Each group will have 25 patients.

Pre-Study Measurements Both groups will have HbA1c measured at the pre-study clinic visit or hospital admission as part of standard of care. After consenting to participation, each subject will schedule a brief telephone check-in with an investigator within 1 week of the initial encounter. Successful adherence to this telephone appointment will be used as a barometer of ability to follow through on scheduled remote communications, and will be required for randomization. After completing the telephone check-in, each patient will return within 2 weeks of the initial encounter. At this visit, randomization will occur, and they will complete 2 questionnaires at the beginning of the study: one knowledge assessment (the Diabetes Knowledge Test 2 (DKT2)) [15] and one assessment of self-efficacy (the Self-Management of Type 1 Diabetes in Adolescence (SMOD-A)) [16].

Intervention Groups Group A will be taught the remote monitoring expectations and will receive training on how to use the Vivify RPM software at the same visit that randomization occurs. Subjects in this group will be enrolled in the RPM protocol for the first 12 weeks of their participation in the study. While on the RPM protocol, subjects will be required to complete the Care Plan questions on a daily basis. They will also have scheduled video conferences with study team physicians or advanced practice nurses on a weekly basis, and will be expected to upload their blood glucose readings to Glooko each week for review. A web-based provider dashboard will allow the study team to monitor patients' usage of the software on a daily basis. Video visits are anticipated to last 15-20 minutes. During this time the study team will review the data collected during the previous week, discuss ongoing diabetes management and any barriers to care, and review selected diabetes self-management educational topics with study participants. The Care Plan questions, Weekly Conference questions, and Educational Objectives intended to be covered during the video visits are appended to the end of this document. Patients in Group B will complete all pre-study measurements at randomization, but remain on a quarterly visit schedule as per standard of care for the first 12 weeks of their participation in the study.

After the first 12 weeks, patients in Group A will return to quarterly office visits with their endocrinology team as per standard of care while patients in Group B enter into the RPM protocol. Both groups will have a clinic visit with HbA1c checked, and will complete the DKT2 and SMOD-A questionnaires for the 2nd time.

The study will conclude with the 6 month visit for both groups. Both groups will have a HbA1c checked, and will complete the post-study DKT2 and SMOD-A questionnaires for the 3rd and final time.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-18 years old
* Diagnosed with Type 1 Diabetes Mellitus >1 year ago with at least one positive diabetes autoantibody
* Patient on multiple daily injections of insulin, with no change to insulin type within the past 3 months
* ≥2 separate HbA1c values (at least 60 days apart) ≥10.0% in the past year, with the most recent HbA1c value ≥10.0%
* English-Speaking (patient and at least 1 parent)
* Patient or parents must own a smart phone or other device compatible with Glooko

Exclusion Criteria:

* Patients on Continuous Subcutaneous Insulin Infusion
* Diagnosed with Type 2 Diabetes or taking metformin
* Other chronic medical condition that would be likely to affect blood glucose. Exceptions include:

  * Hypothyroidism on treatment with normal thyroid function tests
  * Asthma with no oral steroids within past 3 months
* Unstable social situation that could compromise diabetes management or study follow-up in the judgment of the investigators

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 3 months
  To determine whether 12 weeks of participation in a remote monitoring protocol utilizing remote glucose data uploads and video visits through a mobile device improves glycemic control as measured by Hemoglobin A1c in adolescents with poorly controlled Type 1 Diabetes.

SECONDARY OUTCOMES:
Diabetes Knowledge Test 2 (DKT2) score | 6 months
  To determine whether 12 weeks of participation in a remote monitoring protocol can improve diabetes knowledge as assessed by a questionnaire in adolescents with poorly controlled Type 1 Diabetes.
  The DKT2 contains 2 sections, with 23 questions total. The first section is general knowledge, and has 14 items. The second section is an insulin-use subscale, with 9 items. Higher scores are better for both sections.
Self-Management of Type 1 Diabetes in Adolescence (SMOD-A) score | 6 months
  Scoring:
  The first subscale (items 1-13) is Collaboration with Parents. Items 2 and 3 are reversed scored. The range of scores is 0 to 39. Higher scores indicate more collaboration.
  The second subscale is Diabetes Care Activities (items 14-28). Items 16, 21, 22, 23, 25, 26 are reversed scored. The range is 0 to 45. Higher scores indicate better performance of diabetes tasks.
  The third subscale is Diabetes Problem-Solving (items 29-35). Range of scores is 0 to 21. Higher scores indicate better problem-solving.
  The fourth subscale is Diabetes Communication (items 36-45). The range of scores is 0 to 30. Higher scores indicate more communication.
  The fifth subscale, Goals, is composed of items 1-7 of Part II of the instrument. The range of scores is 0 to 21. Higher scores indicate more goals.
  Calculating a total score is not recommended.
DKA Admission Rates | 6 months
  To evaluate whether usage of the remote monitoring protocol affects hospital admission rates for adolescents with poorly controlled Type 1 Diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Soumya Adhikari, MD, Principal Investigator — UT Southwestern
Locations (1):
- Children's Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egro FM. Why is type 1 diabetes increasing? J Mol Endocrinol. 2013 Jul 12;51(1):R1-13. doi: 10.1530/JME-13-0067. Print 2013. PMID 23733895
- [Background] Centers for Disease Control and Prevention., National Diabetes Statistics Report: Estimates of Diabetes and its Burden in the United States, 2014. US Department of Health and Human Services; 2014: Atlanta, GA.
- [Background] Nathan DM; DCCT/EDIC Research Group. The diabetes control and complications trial/epidemiology of diabetes interventions and complications study at 30 years: overview. Diabetes Care. 2014;37(1):9-16. doi: 10.2337/dc13-2112. PMID 24356592
- [Background] Wood JR, Miller KM, Maahs DM, Beck RW, DiMeglio LA, Libman IM, Quinn M, Tamborlane WV, Woerner SE; T1D Exchange Clinic Network. Most youth with type 1 diabetes in the T1D Exchange Clinic Registry do not meet American Diabetes Association or International Society for Pediatric and Adolescent Diabetes clinical guidelines. Diabetes Care. 2013 Jul;36(7):2035-7. doi: 10.2337/dc12-1959. Epub 2013 Jan 22. PMID 23340893
- [Background] Randall L, Begovic J, Hudson M, Smiley D, Peng L, Pitre N, Umpierrez D, Umpierrez G. Recurrent diabetic ketoacidosis in inner-city minority patients: behavioral, socioeconomic, and psychosocial factors. Diabetes Care. 2011 Sep;34(9):1891-6. doi: 10.2337/dc11-0701. Epub 2011 Jul 20. PMID 21775761
- [Background] Ozcan S, Amiel SA, Rogers H, Choudhary P, Cox A, de Zoysa N, Hopkins D, Forbes A. Poorer glycaemic control in type 1 diabetes is associated with reduced self-management and poorer perceived health: a cross-sectional study. Diabetes Res Clin Pract. 2014 Oct;106(1):35-41. doi: 10.1016/j.diabres.2014.07.023. Epub 2014 Jul 26. PMID 25128266
- [Background] Ziegler R, Heidtmann B, Hilgard D, Hofer S, Rosenbauer J, Holl R; DPV-Wiss-Initiative. Frequency of SMBG correlates with HbA1c and acute complications in children and adolescents with type 1 diabetes. Pediatr Diabetes. 2011 Feb;12(1):11-7. doi: 10.1111/j.1399-5448.2010.00650.x. PMID 20337978
- [Background] Campbell MS, Schatz DA, Chen V, Wong JC, Steck A, Tamborlane WV, Smith J, Beck RW, Cengiz E, Laffel LM, Miller KM, Haller MJ; T1D Exchange Clinic Network. A contrast between children and adolescents with excellent and poor control: the T1D Exchange clinic registry experience. Pediatr Diabetes. 2014 Mar;15(2):110-7. doi: 10.1111/pedi.12067. Epub 2013 Aug 19. PMID 23957219
- [Background] Pimouguet C, Le Goff M, Thiebaut R, Dartigues JF, Helmer C. Effectiveness of disease-management programs for improving diabetes care: a meta-analysis. CMAJ. 2011 Feb 8;183(2):E115-27. doi: 10.1503/cmaj.091786. Epub 2010 Dec 13. PMID 21149524
- [Background] Shea S, Weinstock RS, Teresi JA, Palmas W, Starren J, Cimino JJ, Lai AM, Field L, Morin PC, Goland R, Izquierdo RE, Ebner S, Silver S, Petkova E, Kong J, Eimicke JP; IDEATel Consortium. A randomized trial comparing telemedicine case management with usual care in older, ethnically diverse, medically underserved patients with diabetes mellitus: 5 year results of the IDEATel study. J Am Med Inform Assoc. 2009 Jul-Aug;16(4):446-56. doi: 10.1197/jamia.M3157. Epub 2009 Apr 23. PMID 19390093
- [Background] Nundy S, Mishra A, Hogan P, Lee SM, Solomon MC, Peek ME. How do mobile phone diabetes programs drive behavior change? Evidence from a mixed methods observational cohort study. Diabetes Educ. 2014 Nov-Dec;40(6):806-19. doi: 10.1177/0145721714551992. Epub 2014 Oct 2. PMID 25278512
- [Background] Franklin VL, Waller A, Pagliari C, Greene SA. A randomized controlled trial of Sweet Talk, a text-messaging system to support young people with diabetes. Diabet Med. 2006 Dec;23(12):1332-8. doi: 10.1111/j.1464-5491.2006.01989.x. PMID 17116184
- [Background] Malloy LE, Gingerich J, Olson MD, Atkins DL. Remote monitoring of cardiovascular implantable devices in the pediatric population improves detection of adverse events. Pediatr Cardiol. 2014 Feb;35(2):301-6. doi: 10.1007/s00246-013-0774-5. Epub 2013 Aug 15. PMID 23949666
- [Background] Jacob E, Duran J, Stinson J, Lewis MA, Zeltzer L. Remote monitoring of pain and symptoms using wireless technology in children and adolescents with sickle cell disease. J Am Assoc Nurse Pract. 2013 Jan;25(1):42-54. doi: 10.1111/j.1745-7599.2012.00754.x. Epub 2012 Jul 12. PMID 23279278
- [Result] Fitzgerald JT, Funnell MM, Anderson RM, Nwankwo R, Stansfield RB, Piatt GA. Validation of the Revised Brief Diabetes Knowledge Test (DKT2). Diabetes Educ. 2016 Apr;42(2):178-87. doi: 10.1177/0145721715624968. Epub 2016 Jan 14. PMID 26769757
- [Result] Schilling LS, Dixon JK, Knafl KA, Lynn MR, Murphy K, Dumser S, Grey M. A new self-report measure of self-management of type 1 diabetes for adolescents. Nurs Res. 2009 Jul-Aug;58(4):228-36. doi: 10.1097/NNR.0b013e3181ac142a. PMID 19561555